CLINICAL TRIAL: NCT01893268
Title: Therapeutic Strategies Including Avastin as 1st Line Therapy in Elderly Patients Suffering From Advanced (IIIB/IV Stage) Non-squamous Non-small Cell Lung Cancer, in Routine Clinical Practice.
Brief Title: An Observational Study of Avastin (Bevacizumab) in Elderly Patients With Non-Squamous Non-Small Cell Lung Cancer in Clinical Practice
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28621
Record Dates: First submitted 2013-07-02; First posted 2013-07-08 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This prospective, observational study will assess the effectiveness and safety of Avastin (bevacizumab) as 1st line therapy in elderly patients with advanced non-squamous non-small cell lung cancer in clinical practice. Therapy with Avastin and standard chemotherapy will be administered according to the treating physician. Data will be collected for approximately 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >= 65 years of age
* Diagnosis of advanced non squamous Non-Small Cell Lung Carcinoma (nsNSCLC, stage IIIB or IV) for whom the physician has decided to initiate a treatment with Avastin combined with chemotherapy as 1st line therapy
* Having received oral and written information about the study, and having signed a written consent form

Exclusion Criteria:

* Participation in a cancer clinical trial with an investigational medicinal product other than this study
* Patient previously treated with Avastin
* Patient under supervision or guardianship

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged over 65 years with non-squamous non-small cell lung cancer
Sampling Method: Probability Sample
Enrollment: 279 (Actual)
Dates: Start 2013-07-25 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2018-03-20 (Actual)

PRIMARY OUTCOMES:
Proportion of patients treated with a chemotherapy in combination with Avastin including description of chemotherapy regimens and management of Avastin treatment | Approximately 4 years

SECONDARY OUTCOMES:
Characteristics of patients with advanced non-squamous non-small cell lung cancer | Approximately 4 years
Tumor characteristics of patients with advanced non-squamous non-small cell lung cancer | Approximately 4 years
Progression-free survival | Approximately 4 years
Overall survival | Approximately 4 years
Quality of Life | Approximately 4 years
Safety: Incidence of adverse events | Approximately 4 years
Reasons of non-use of Avastin as first-line therapy | Approximately 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (88):
- France (88):
  - Clinique Du Docteur Calabet; Cromg, Agen
  - Ch Du Pays D Aix; Pneumologie, Aix-en-Provence
  - Poly Parc Rambot La Provencale; Chimiotherapie Ambulatoire, Aix-en-Provence
  - Cabinet Medical, Amiens
  - Centre Hospitalier Uni Ire; Pneumology, Angers
  - Chic Cote Basque Bayonne; Pneumologie, Bayonne
  - HOPITAL JEAN MINJOZ; Oncologie, Besançon
  - CH Germon ET Gauthier; Pneumologie, Beuvry
  - Ch De Beziers; Pneumologie, Béziers
  - Hopital Avicenne; Cancerologie, Bobigny
  - Polyclinique Bordeaux Nord Aquitaine; Chimiotherapie Radiotherapie, Bordeaux
  - Centre Hospitalier Fleyriat; Oncologie/Hematologie, Bourg-en-Bresse
  - Ch De Fleyriat; Pneumologie 1, Bourg-en-Bresse
  - Hia Clermont Tonnerre; Pneumologie, Brest
  - Ch De Brive La Gaillarde; Radiotherapie Oncologie, Brive-la-Gaillarde
  - Hopital Louis Pradel; Pneumologie, Bron
  - Hopital Pierre Nouveau; Pneumologie, Cannes
  - Ch Antoine Gayraud; Oncologie, Carcassonne
  - Clinique Du Parc; Hematologie, Castelnau Lez
  - Ctre Medical Nicolas de Pontoux, Chalon-sur-Saône
  - Ch De Chauny; Pneumologie, Chauny
  - CH Du Cotentin Site De Cherbourg; Hopital De Jour, Cherbourg Octeville
  - Hopital Gabriel Montpied; Service de Pneumologie, Clermont-Ferrand
  - Centre Jean Perrin; Hopital De Semaine, Clermont-Ferrand
  - Hopital Louis Pasteur; Pneumologie Tabacologie, Colmar
  - Centre Hospitalier Alpes Leman CHAL;Pneumologie, Contamine-sur-Arve
  - Clinique Des Cedres; Pneumologie, Cornebarrieu
  - Centre Hospitalier Intercommunal; Service de Pneumologie, Créteil
  - Chu Site Du Bocage;Pneumologie, Dijon
  - Ch De La Dracenie; Pneumologie, Draguignan
  - Centre D Oncologie Dunkerquois, Dunkirk
  - Chi Emile Durkheim Site Epinal; Pneumologie, Épinal
  - Chi Alpes Du Sud Site De Gap; Pneumologie, Gap
  - Hopital Nord Ouest;Unite 2c, Gleizé
  - CH Emmanuel Rain; Oncologie, Gonesse
  - Hopital Prive De Chantilly; Medecine, Gouvieux Chantilly
  - Hopital D Hayange;Medecine A Et P, Hyères
  - Centre Oscar Lambret; Chir Cancerologie General, Lille
  - Hopital Saint Vincent; Consult et Explorations, Lille
  - Hopital Calmette; Pneumologie Oncologie Ouest, Lille
  - Clinique Chenieux; Oncology, Limoges
  - Hopital Du Cluzeau; Service de Pathologie Respiratoire, Limoges
  - Hopital Dupuytren; Pneumologie, Limoges
  - Centre Hospitalier Général; Pneumologie, Longjumeau
  - Ch Bretagne Sud Site Scorff; Oncologie Medicale, Lorient
  - Centre Medical Parot, Lyon
  - Centre Hospitalier François Quesnay; Pneumologie-Neurologie, Mantes-la-Jolie
  - Hôpital Saint Joseph; Oncologie Medicale, Marseille
  - Centre Hospitalier; Pneumologie, Metz-Tessy
  - Hopital Layne; Medecine Ambulatoire, Mont-de-Marsan
  - Ch De Montauban; Pneumologie, Montauban
  - Hopital Emile Muller;Pneumologie, Mulhouse
  - Cabinet Medical, Nancy
  - Polyclinique Gentilly; CHIMIOTHERAPIE AMBULATOIRE, Nancy
  - Hopital Caremeau; Pneumologie, Nîmes
  - Clinique sainte marie; chimiotherapie ambulatoire, Osny
  - Hopital Cochin; Unite Fonctionnelle D Oncologie, Paris
  - Hopital Saint Louis; Oncologie Medicale, Paris
  - Hopital Europeen Georges Pompidou; Service D'Oncologie Medicale, Paris
  - Centre Catalan D' Oncologie, Perpignan
  - Centre Hospitalier Lyon Sud; Pneumologie, Pierre-Bénite
  - CH Rene Dubos; Oncologie, Pontoise
  - Hopital Laennec; Service de Pneumologie, Quimper
  - Ch De Rambouillet; Pneumologie Cardiologie, Rambouillet
  - Cabinet, Reims
  - Hopital de Pontchaillou; Service de Pneumologie, Rennes
  - Clinique Saint Hilaire; Sce Chimiotherapie, Rouen
  - Centre Cardiologique Du Nord; Pneumologie, Saint-Denis
  - Clinique de L'Union; Oncologie, Saint-Jean
  - Cabinet Medical, Saint-Laurent-du-Var
  - Hopital Nord; Service de Pneumologie, Saint-Priest-en-Jarez
  - Ch De Saint Quentin; Medecine B14, Saint-Quentin
  - Ch De Saintonge; Unite 2 Pneumologie, Saintes
  - Centre Medical National Mgen; Pneumologie, Ste Feyre
  - Centre Paul Strauss; Oncologie Medicale, Strasbourg
  - Hopital Bel Air; Pneumologie Allergologie, Thionville
  - Hopitaux Du Leman Site Thonon; Pneumologie, Thonon-les-Bains
  - Hia Sainte Anne; Pneumologie, Toulon
  - Hopital Sainte Musse; Pneumologie, Toulon
  - Clinique Pasteur; Pneumologie, Toulouse
  - Groupe Oncorad Garonne; Unite Onco Hematologie, Toulouse
  - Cabinet Medical, Tours
  - Hopital Des Hauts Clos; Pneumologie, Troyes
  - Ch De Valence; Medecine 7, Valence
  - Centre Alexis Vautrin; Oncologie Medicale, Vandœuvre-lès-Nancy
  - Hopital Robert Schuman; Pneumologie, Vantoux
  - Hopital Saint Nicolas; Pneumologie, Verdun
  - Gh Mutualiste Les Portes Du Sud; Pneumologie, Vénissieux